CLINICAL TRIAL: NCT06804213
Title: A Randomized Controlled Study Evaluating Student Wellness Using the Roadmap mHealth App and Wellness Coaching
Brief Title: Student Wellness 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: STEER for Student Athletes (Unknown)
Responsible Party: Principal Investigator, Sung Won Choi, Edith S Briskin and Shirley K Schlafer Foundation Research Professor of Pediatrics and Associate Professor of Pediatrics and Communicable Diseases, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00257823
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Issue
Keywords: mobile health; wearable sensors; college students; wellness coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wellness coaching plus mobile health app (positive activities) (Experimental): Participants will participate in wellness coaching and receive a wearable device, and they will be assigned to use the mobile health app with positive psychological activities installed. Additionally, participants can view their daily step count and number of hours of sleep in the mobile health app.
  Interventions: Behavioral: Mobile health app with positive psychological activities
- Wellness coaching plus limited mobile health app (no positive activities) (No Intervention): Participants will participate in wellness coaching and receive a wearable device, but will be assigned to use the mobile health app WITHOUT positive psychological activities installed. Participants can only view their daily step count and number of hours of sleep in the mobile health app.

INTERVENTIONS:
Behavioral: Mobile health app with positive psychological activities — Mobile health app with step tracking, sleep tracking, and positive psychological activities
  Arms: Wellness coaching plus mobile health app (positive activities)

SUMMARY:
In this randomized controlled study, investigators plan to assess the impact of a mobile health app with positive psychological combined with wellness coaching on college student mental health outcomes. The study aims to differentiate the effectiveness of combining mobile health and wellness coaching compared to wellness coaching on its own. The goal is to improve our understanding of the optimal combination of traditional in-person and digital interventions on diverse student populations, as well as better understand the causal impact of the mobile health app on well-being.

DETAILED DESCRIPTION:
Study participants will be asked to:

1. Complete as many sessions of individual wellness coaching as they see fit
2. Install and interact with the Fitbit and Roadmap 2.0 apps on their smartphone
3. Complete longitudinal surveys at baseline, month 1, month 2, and end of study
4. Complete an exit interview at the end of the study

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years old.
2. Students must be either enrolled at the University of Michigan OR in the STEER transition program.
3. Potential subjects must be able to provide a mailing address within the United States where they can receive study tools and be mailed study materials (e.g., Fitbit, compensation).
4. Possess a smartphone (Apple or Android).
5. Ability to understand and demonstrate willingness to remotely sign a written informed consent document

Exclusion Criteria:

1. People who are not enrolled in classes at the University of Michigan OR people who are not members of the STEER organization.
2. Unwilling or unable to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of Roadmap 2.0 plus wellness coaching on college student mental health | From enrollment to the exit survey at 4 months
  Evaluate the difference between the intervention (Roadmap 2.0 + wellness coaching) arm and the control (limited Roadmap 2.0 + wellness coaching) arm by measuring the effectiveness of Roadmap 2.0 when coupled with wellness coaching. Participants will complete validated quality-of-life surveys, which measure subject-reported outcomes related to mental health.

SECONDARY OUTCOMES:
Survey completion | From enrollment to the exit survey at 4 months
  Assess survey completion rate, estimating at least 50% of participants will complete the surveys at all four time points.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - STEER for Student Athletes, Port Chester, New York

IPD SHARING:
Plan to Share IPD: No